CLINICAL TRIAL: NCT05184192
Title: Efficacy of Gabapentin for Post-Covid-19 Olfactory Dysfunction
Acronym: GRACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202110011
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; Olfactory Disorder; Anosmia; Hyposmia; Parosmia
MeSH Terms: conditions — COVID-19; Anosmia; Olfaction Disorders

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded, both participants and investigators will be blinded. Intervention will be packaged in blinded fashion by pharmacist before being shipped to participants by research assistant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): This arm will be given the active treatment, oral Letco (gabapentin) gelatin capsules of 300mg each.
  Up to the first four weeks will be a titration period (week 1 300mg TID, week 2 600mg TID, week 3 900mg TID, week 4 1,200mg TID) as tolerated. If intolerable adverse reactions occur, the dosage will be decreased to prior tolerable dose (e.g., if 900mg TID is intolerable, dose will be decreased to 600mg TID).
  The following eight weeks will be fixed dose, the highest tolerable dose from the titration period.
  Up to two weeks will be a taper down tailored to the maximum dose the participant reached during the titration and fixed periods.
  A maximum 14 weeks will mark the end of active treatment. Follow-up assessments will be conducted 4 weeks after completion of the taper-down period.
  Interventions: Drug: Gabapentin gelatin capsules 300mg
- Placebo (Placebo Comparator): Placebo gelatin capsules that look, smell, and taste like gabapentin capsules will be given to the placebo arm.
  To preserve double-blinding of the study, subjects will receive one capsule TID the first week, the second week two capsules TID, the third week three capsules TID, and fourth week four capsules TID as tolerated. If intolerable, the dose will be decreased to prior tolerable dose.
  The next eight weeks will be a fixed amount of placebo based on the highest tolerable amount from the titration period.
  Subjects will then taper-down placebo to imitate the gabapentin arm for maximum two weeks based on highest dose achieved during study.
  4 weeks after completion of taper-down, follow-up assessments will be conducted.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin gelatin capsules 300mg — Gabapentin is an anti-epileptic also used for nerve pain. This study will investigate the efficacy of gabapentin for olfactory nerve recovery and improvement in post-Covid-19 olfactory dysfunction.
  Other Names: Letco
  Arms: Gabapentin
Drug: Placebo — lactose monohydrate NF
  Arms: Placebo

SUMMARY:
This study will investigate the efficacy of oral gabapentin in olfactory improvement following Covid-19- associated olfactory dysfunction. This is a randomized, double-blinded, placebo-controlled trial.

DETAILED DESCRIPTION:
The drug will be given over a maximum 14 weeks with up to four weeks titrating up, eight weeks maintaining highest tolerable dose, and up to two weeks tapering down. Change in olfactory function from baseline to completion of 8-week fixed-dose period will be compared between the two study groups. Follow-up assessments will be conducted for both groups 4 weeks after completion of taper down.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years
* Residing within the states of Missouri or Illinois
* Clinically diagnosed or subjective olfactory dysfunction (anosmia, hyposmia, or parosmia) of 3 months duration or longer diagnosed within 2 weeks of Covid-19 infection
* UPSIT score consistent with diminished olfactory function (score ≤ 33 in men and ≤ 34 in women).
* Willing to respond daily to study surveys, preferably through smartphone with unlimited texting plan
* In possession of ALL 7 household items: soap, burnt candle, peanut butter, herb, garlic, lemon, and coffee

Exclusion Criteria:

* Clinically diagnosed olfactory dysfunction secondary to genetic abnormalities or congenital dysfunction, trauma, non-Covid-19 viral infection, nasal polyps, neurodegenerative disorders
* Current use of: azelastine, bromperidol, orophenadrine, oxomemazine, kratom, paraldehyde, or thalidomide
* History of addiction to alcohol, cocaine, or opioids
* Impaired renal function, myasthenia gravis, or myoclonus
* Severe allergy to peanuts
* Pregnancy or attempting pregnancy during study participation
* Inability to participate in virtual trial due to lack of access to the internet or unlimited text messaging; inability to comprehend or use English language
* Availability less than 6 months from time of enrollment
* Residency in states other than Missouri or Illinois.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Background] Boscolo-Rizzo P, Borsetto D, Fabbris C, Spinato G, Frezza D, Menegaldo A, Mularoni F, Gaudioso P, Cazzador D, Marciani S, Frasconi S, Ferraro M, Berro C, Varago C, Nicolai P, Tirelli G, Da Mosto MC, Obholzer R, Rigoli R, Polesel J, Hopkins C. Evolution of Altered Sense of Smell or Taste in Patients With Mildly Symptomatic COVID-19. JAMA Otolaryngol Head Neck Surg. 2020 Aug 1;146(8):729-732. doi: 10.1001/jamaoto.2020.1379. PMID 32614442
- [Background] Hummel T, Rissom K, Reden J, Hahner A, Weidenbecher M, Huttenbrink KB. Effects of olfactory training in patients with olfactory loss. Laryngoscope. 2009 Mar;119(3):496-9. doi: 10.1002/lary.20101. PMID 19235739
- [Background] Turner JH. Olfactory training: what is the evidence? Int Forum Allergy Rhinol. 2020 Nov;10(11):1199-1200. doi: 10.1002/alr.22681. Epub 2020 Sep 3. No abstract available. PMID 32776673
- [Background] Biole C, Bianco M, Nunez-Gil IJ, Cerrato E, Spirito A, Roubin SR, Viana-Llamas MC, Gonzalez A, Castro-Mejia AF, Eid CM, Fernandez-Perez C, Uribarri A, Alfonso-Rodriguez E, Ugo F, Guerra F, Feltes G, Akin I, Fernandez-Rozas I, Blasco-Angulo N, Huang J, Aguado MG, Pepe M, Romero R, Becerra-Munoz VM, Estrada V, Macaya C. Gender Differences in the Presentation and Outcomes of Hospitalized Patients With COVID-19. J Hosp Med. 2021 Jun;16(6):349-352. doi: 10.12788/jhm.3594. PMID 34129486
- [Background] Butowt R, von Bartheld CS. Anosmia in COVID-19: Underlying Mechanisms and Assessment of an Olfactory Route to Brain Infection. Neuroscientist. 2021 Dec;27(6):582-603. doi: 10.1177/1073858420956905. Epub 2020 Sep 11. PMID 32914699
- [Background] Bilinska K, Butowt R. Anosmia in COVID-19: A Bumpy Road to Establishing a Cellular Mechanism. ACS Chem Neurosci. 2020 Aug 5;11(15):2152-2155. doi: 10.1021/acschemneuro.0c00406. Epub 2020 Jul 16. PMID 32673476
- [Background] Kuba K, Imai Y, Penninger JM. Multiple functions of angiotensin-converting enzyme 2 and its relevance in cardiovascular diseases. Circ J. 2013;77(2):301-8. doi: 10.1253/circj.cj-12-1544. Epub 2013 Jan 18. PMID 23328447
- [Background] Mollica V, Rizzo A, Massari F. The pivotal role of TMPRSS2 in coronavirus disease 2019 and prostate cancer. Future Oncol. 2020 Sep;16(27):2029-2033. doi: 10.2217/fon-2020-0571. Epub 2020 Jul 13. No abstract available. PMID 32658591
- [Background] Damm M, Pikart LK, Reimann H, Burkert S, Goktas O, Haxel B, Frey S, Charalampakis I, Beule A, Renner B, Hummel T, Huttenbrink KB. Olfactory training is helpful in postinfectious olfactory loss: a randomized, controlled, multicenter study. Laryngoscope. 2014 Apr;124(4):826-31. doi: 10.1002/lary.24340. Epub 2013 Sep 19. PMID 23929687
- [Background] Schopf CL, Ablinger C, Geisler SM, Stanika RI, Campiglio M, Kaufmann WA, Nimmervoll B, Schlick B, Brockhaus J, Missler M, Shigemoto R, Obermair GJ. Presynaptic alpha2delta subunits are key organizers of glutamatergic synapses. Proc Natl Acad Sci U S A. 2021 Apr 6;118(14):e1920827118. doi: 10.1073/pnas.1920827118. PMID 33782113
- [Background] Lopez-D'alessandro E, Escovich L. Combination of alpha lipoic acid and gabapentin, its efficacy in the treatment of Burning Mouth Syndrome: a randomized, double-blind, placebo controlled trial. Med Oral Patol Oral Cir Bucal. 2011 Aug 1;16(5):e635-40. doi: 10.4317/medoral.16942. PMID 20711135
- [Background] Doty RL, Shaman P, Kimmelman CP, Dann MS. University of Pennsylvania Smell Identification Test: a rapid quantitative olfactory function test for the clinic. Laryngoscope. 1984 Feb;94(2 Pt 1):176-8. doi: 10.1288/00005537-198402000-00004. PMID 6694486
- [Background] Doty RL. Olfactory dysfunction and its measurement in the clinic. World J Otorhinolaryngol Head Neck Surg. 2015 Oct 26;1(1):28-33. doi: 10.1016/j.wjorl.2015.09.007. eCollection 2015 Sep. PMID 29204537
- [Background] Mersfelder TL, Nichols WH. Gabapentin: Abuse, Dependence, and Withdrawal. Ann Pharmacother. 2016 Mar;50(3):229-33. doi: 10.1177/1060028015620800. Epub 2015 Dec 31. PMID 26721643
- [Derived] Mahadev A, Hentati F, Miller B, Bao J, Perrin A, Kallogjeri D, Piccirillo JF. Efficacy of Gabapentin For Post-COVID-19 Olfactory Dysfunction: The GRACE Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Dec 1;149(12):1111-1119. doi: 10.1001/jamaoto.2023.2958. PMID 37733356
- See also: World Health Organization Covid-19 Dashboard — http://covid19.who.int/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: This arm will be given the active treatment, oral Letco (gabapentin) gelatin capsules of 300mg each.
  Up to the first four weeks will be a titration period (week 1 300mg TID, week 2 600mg TID, week 3 900mg TID, week 4 1,200mg TID) as tolerated. If intolerable adverse reactions occur, the dosage will be decreased to prior tolerable dose (e.g., if 900mg TID is intolerable, dose will be decreased to 600mg TID).
  The following eight weeks will be fixed dose, the highest tolerable dose from the titration period.
  Up to two weeks will be a taper down tailored to the maximum dose the participant reached during the titration and fixed periods.
  A maximum 14 weeks will mark the end of active treatment. Follow-up assessments will be conducted 4 weeks after completion of the taper-down period.
  Gabapentin gelatin capsules 300mg: Gabapentin is an anti-epileptic also used for nerve pain. This study will investigate the efficacy of gabapentin for olfactory nerve recovery and improvement in post-Covid-19 olfactory dysfunction.
- Placebo: Placebo gelatin capsules that look, smell, and taste like gabapentin capsules will be given to the placebo arm.
  To preserve double-blinding of the study, subjects will receive one capsule TID the first week, the second week two capsules TID, the third week three capsules TID, and fourth week four capsules TID as tolerated. If intolerable, the dose will be decreased to prior tolerable dose.
  The next eight weeks will be a fixed amount of placebo based on the highest tolerable amount from the titration period.
  Subjects will then taper-down placebo to imitate the gabapentin arm for maximum two weeks based on highest dose achieved during study.
  4 weeks after completion of taper-down, follow-up assessments will be conducted.
  Placebo: lactose monohydrate NF
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 34 | 34
Completed | 26 | 17
Not Completed | 8 | 17
Not completed — Lost to Follow-up | 4 | 7
Not completed — Adverse Event | 1 | 4
Not completed — PI withdrawal | 1 | 2
Not completed — Withdrew due to adverse effect | 1 | 0
Not completed — Medication schedule | 1 | 0
Not completed — Concern for adverse effects | 0 | 4

BASELINE CHARACTERISTICS:
Population: Thirty-four participants were randomized to gabapentin and 34 were randomized to placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10.6) | 44 (15.5) | 43 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Seven participants withdrew prior to baseline survey completion.
  Participants
    number analyzed (Participants) | 27 | 34 | 61
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 23 | 33 | 56
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 7 participants withdrew prior to the baseline survey completion.
  Participants
    White: number analyzed (Participants) | 27 | 34 | 61
    White | 23 | 33 | 56
    Black / African American: number analyzed (Participants) | 27 | 34 | 61
    Black / African American | 2 | 0 | 2
    Hispanic: number analyzed (Participants) | 27 | 34 | 61
    Hispanic | 0 | 1 | 1
    Other: number analyzed (Participants) | 27 | 34 | 61
    Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68
University of Pennsylvania Smell Identification Test (UPSIT) [Median (Full Range); unit: score on a scale (0-40)] — Forty different odors are presented in this test. Scoring: Forced choice of 4 responses to identify each smell. Anosmia: score 6-18; severe microsmia: score 19-25, moderate microsmia: 26-30 in women and 26-29 in men; mild microsmia: 31-34 in women and 30-33 in men; and normosmia: score > 34 in women and >33 in men.
  The total UPSIT score can range from 0 to 40 and scores. The MCID in UPSIT score is 4. Population: Seven participants withdrew prior to baseline survey completion.
  score on a scale (0-40)
    number analyzed (Participants) | 27 | 34 | 61
    (all) | 24.5 [8 to 33] | 25.5 [7 to 34] | 25.0 [7.0 to 34.0]
Olfactory Dysfunction Outcomes Rating (ODOR) [Median (Full Range); unit: score on a scale (0-112)] — Olfactory Dysfunction Outcomes Rating (ODOR). The ODOR questionnaire is a 28-item disease-specific health status survey to assess the physical problems, functional impairments, and emotional consequences secondary to olfactory dysfunction.
  Results The ODOR is a 28-item instrument with each item scored as either no difficulty or very rarely bothered (0) to complete difficulty or very frequently bothered (4) with a total instrument score range of 0 to 112 points. Higher scores indicate higher degree of dysfunction and limitation
  The MCID is 15. Population: Seven participants withdrew prior to baseline survey completion.
  score on a scale (0-112)
    number analyzed (Participants) | 27 | 34 | 61
    (all) | 56 [14 to 102] | 54.5 [0 to 101] | 56 [0 to 102]
NASAL-7 categories [Count of Participants; unit: Participants] — Seven participants withdrew prior to baseline survey completion. Population: 7 patients were excluded and not analyzed as previously explained.
  Participants
    Anosmia (0-4): number analyzed (Participants) | 27 | 34 | 61
    Anosmia (0-4) | 9 | 11 | 20
    Severe dysfunction (5-7): number analyzed (Participants) | 27 | 34 | 61
    Severe dysfunction (5-7) | 12 | 16 | 28
    Mild dysfunction (8-10): number analyzed (Participants) | 27 | 34 | 61
    Mild dysfunction (8-10) | 4 | 5 | 9
    Normosmia (11-14): number analyzed (Participants) | 27 | 34 | 61
    Normosmia (11-14) | 2 | 2 | 4
CGI-S of smell [Count of Participants; unit: Participants] — The CGI-Severity scale ranges from 1 to 7, where 1 is normal function and 7 is complete anosmia. This assessment will provide subjective data on patients' baseline olfactory function prior to beginning the trial, after 8-week Fixed-Dose period, and 4 weeks after completion of Taper-Down phase. Population: 7 participants withdrew prior to the baseline survey completion.
  Participants
    Absent: number analyzed (Participants) | 27 | 34 | 61
    Absent | 6 | 5 | 11
    Poor: number analyzed (Participants) | 27 | 34 | 61
    Poor | 17 | 20 | 37
    Fair: number analyzed (Participants) | 27 | 34 | 61
    Fair | 3 | 7 | 10
    Good: number analyzed (Participants) | 27 | 34 | 61
    Good | 1 | 1 | 2
    Very good: number analyzed (Participants) | 27 | 34 | 61
    Very good | 0 | 1 | 1
    Excellent: number analyzed (Participants) | 27 | 34 | 61
    Excellent | 0 | 0 | 0
CGI-S of parosmia [Count of Participants; unit: Participants] — Population: Seven participants withdrew prior to baseline survey completion.
  Participants
    Complete distortion: number analyzed (Participants) | 27 | 34 | 61
    Complete distortion | 9 | 9 | 18
    Mostly distorted: number analyzed (Participants) | 27 | 34 | 61
    Mostly distorted | 13 | 10 | 23
    Moderate distortion: number analyzed (Participants) | 27 | 34 | 61
    Moderate distortion | 5 | 9 | 14
    Mild distortion: number analyzed (Participants) | 27 | 34 | 61
    Mild distortion | 0 | 4 | 4
    No distortion: number analyzed (Participants) | 27 | 34 | 61
    No distortion | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression of Improvement Scale (CGI-I)
Description: The primary outcome measure was the treatment response rate following the 8-week FD phase as determined by the CGI-I. The CGI-I is a modified 7-point Likert scale of -perceived change.
  Response options include: (1) much better, (2) somewhat better, (3) slightly better), (4) neither better nor worse, (5) slightly worse, (6) somewhat worse, (7) much worse. The response rate was defined as the number of participants self-reporting at least "slightly better" divided by the number of participants in each treatment group. Th
Time Frame: After the 8 week FD phase and four week post-tapper
Population: 26 participants in the placebo group completed the treatment, but 25 participants completed the posttaper survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 32
Participants
  Fixed Dose Period | 8 | 20
  4 week post tapper: number analyzed (Participants) | 16 | 25
  4 week post tapper | 7 | 12

2. Secondary Outcome: University of Pennsylvania Smell Identification Test (UPSIT)
Description: Forty different odors are presented in this test.
  Scoring: Forced choice of 4 responses to identify each smell. Anosmia: score 6-18; severe microsmia: score 19-25, moderate microsmia: 26-30 in women and 26-29 in men; mild microsmia: 31-34 in women and 30-33 in men; and normosmia: score > 34 in women and >33 in men.
  The total UPSIT score can range from 0 to 40 and scores. The MCID in UPSIT score is 4.
  Scores are interpreted as the level of absolute smell function (i.e., normosmia, mild hyposmia, moderate hyposmia, severe hyposmia, and anosmia), using the age- and sex-related normative classification system described in the UPSIT manual (Table 1)
Time Frame: Baseline, after completion of eight-week fixed-dose period, and 4 weeks after completion of taper-down period
Population: 26 participants in placebo group completed treatment, but 25 participants completed the posttaper survey. 18 participants in the gabapentin group completed treatment, but 16 participants completed the post-taper survey.
Measure: Median (Full Range); unit: score on a scale (0-40)
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 26
score on a scale (0-40)
  Baseline | 23 [10 to 31] | 24 [7 to 34]
  Fixed Dose | 25 [12 to 34] | 25 [15 to 34]
  Post-taper: number analyzed (Participants) | 16 | 25
  Post-taper | 26 [7 to 33] | 25 [9 to 35]

3. Secondary Outcome: Olfactory Dysfunction Outcomes Rating (ODOR)
Description: The ODOR questionnaire is a validated 28-item patient-reported outcome measure which assesses the physical, functional, and emotional consequences of OD.
  The ODOR is a 28-item instrument with each item scored as either no difficulty or very rarely bothered (0) to complete difficulty or very frequently bothered (4) with a total instrument score range of 0 to 112 points. Higher scores indicate higher degree of dysfunction and limitation. the MCID is 15 points.
Time Frame: Baseline, after completion of eight-week fixed-dose period, and 4 weeks after completion of taper-down period
Population: 26 participants in placebo group completed treatment, but 25 participants completed the posttaper survey.
  18 participants in the gabapentin group completed treatment, but 16 participants completed the post-taper survey.
  Each of the 28 items is scored 0 to 4. The maximum total score is 112 with higher scores representing greater quality of life impairment.
  The MCID is 15.
Measure: Median (Full Range); unit: score on a scale (0-112)
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 26
score on a scale (0-112)
  Baseline | 23 [10 to 31] | 54.5 [30 to 96]
  Fixed Dose | 25.5 [15 to 34] | 49.9 [8 to 96]
  Post Taper: number analyzed (Participants) | 16 | 25
  Post Taper | 25 [9 to 35] | 45 [8 to 85]

4. Secondary Outcome: NASAL-7
Description: NASAL-7 is a simple diagnostic tool for olfactory dysfunction that is based on commonly found household items and can be used by adults who suspect olfactory dysfunction. The NASAL-7 was developed by Dr. Piccirillo and colleagues in the Clinical Outcomes Research Office. The NASAL-7, contains 7 household items with each item scored as 0 for 'Cannot Smell', 1 for 'Smells Less Strong/Different Than Normal', and 2 for 'Smells Normal', for a total possible score ranging from 0-14. The following four categories of olfactory function were defined based on NASAL-7 score: anosmia (score 0-4), severe dysfunction (score 5-7), mild dysfunction (score 8-10), and normosmia (score 11-14).
Time Frame: Baseline, after completion of eight-week fixed-dose period, and 4 weeks after completion of taper-down period
Population: 26 participants in placebo group completed treatment, but 25 participants completed the posttaper survey. 18 participants in the gabapentin group completed treatment, but 16 participants completed the posttaper survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 26
Participants
  Baseline: Anosmia (0-4) | 6 | 10
  Baseline: Severe dysfunction (5-7) | 8 | 12
  Baseline: Mild dysfunction (8-10) | 2 | 3
  Baseline: Normosmia (11-14) | 2 | 1
  Fixed Dose: Anosmia (0-4) | 4 | 7
  Fixed Dose: Severe dysfunction (5-7) | 5 | 9
  Fixed Dose: Mild dysfunction (8-10) | 4 | 6
  Fixed Dose: Normosmia (11-14) | 5 | 4
  Post taper: number analyzed (Participants) | 16 | 25
  Post taper: Anosmia (0-4) | 5 | 7
  Post taper: Severe dysfunction (5-7) | 6 | 6
  Post taper: Mild dysfunction (8-10) | 2 | 5
  Post taper: Normosmia (11-14) | 3 | 7

5. Secondary Outcome: CGI-Severity of Smell
Description: CGI-Severity. The CGI-Severity scale ranges from 1 to 7, where 1 is normal function and 7 is complete anosmia. This assessment will provide subjective data on patients' baseline olfactory function prior to beginning the trial, after 8-week Fixed-Dose period, and 4 weeks after completion of Taper-Down phase
Time Frame: 8-week Fixed-Dose period, and 4 weeks after completion of Taper-Down phase
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 26
Participants
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Absent | 4 | 4
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Poor | 12 | 16
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Fair | 1 | 4
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Good | 1 | 1
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Very good | 0 | 1
  Assessments of the Secondary Outcome Measures of Study Groups: Baseline: Excellent | 0 | 0
  Fixed Dose: Absent | 3 | 5
  Fixed Dose: Poor | 4 | 13
  Fixed Dose: Fair | 8 | 4
  Fixed Dose: Good | 3 | 3
  Fixed Dose: Very good | 0 | 1
  Fixed Dose: Excellent | 0 | 0
  Post taper: number analyzed (Participants) | 16 | 25
  Post taper: Absent | 2 | 3
  Post taper: Poor | 7 | 13
  Post taper: Fair | 5 | 6
  Post taper: Good | 2 | 2
  Post taper: Very good | 0 | 1
  Post taper: Excellent | 0 | 0

6. Secondary Outcome: CGI-S of Parosmia
Description: Clinical Global Impression-Severity Scale for Parosmics (CGI-P). The CGI-P Scale is a global rating of parosmia and the single global rating ranges from 1-5, where 1 is No Distortion, 2 is Mild Distortion, 3 is Moderate Distortion, 4 is Mostly Distorted, and 5 is Complete Distortion. The response on the CGI-P will provide information on the patient's perceived severity of the distortion of their smell.
Time Frame: 8-week Fixed-Dose period, and 4 weeks after completion of Taper-Down phase
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 18 | 26
Participants
  Assessments of Secondary Outcome Measures of Study Groups: Baseline: Complete Distortion | 7 | 6
  Assessments of Secondary Outcome Measures of Study Groups: Baseline: Mostly Distorted | 9 | 8
  Assessments of Secondary Outcome Measures of Study Groups: Baseline: Moderate Distortion | 2 | 7
  Assessments of Secondary Outcome Measures of Study Groups: Baseline: Mild Distortion | 0 | 4
  Assessments of Secondary Outcome Measures of Study Groups: Baseline: No Distortion | 0 | 1
  Fixed Dose: Complete Distortion | 2 | 3
  Fixed Dose: Mostly Distorted | 6 | 6
  Fixed Dose: Moderate Distortion | 4 | 9
  Fixed Dose: Mild Distortion | 5 | 7
  Fixed Dose: No Distortion | 1 | 1
  Post tapper: number analyzed (Participants) | 16 | 25
  Post tapper: Complete Distortion | 2 | 2
  Post tapper: Mostly Distorted | 5 | 9
  Post tapper: Moderate Distortion | 6 | 9
  Post tapper: Mild Distortion | 2 | 4
  Post tapper: No Distortion | 1 | 1

ADVERSE EVENTS:
Time Frame: If tolerated, all participants will complete the Titration period (≤ 4 weeks), Fixed-Dose period (8 weeks), and Taper-Down period (2 weeks) for maximum 14 weeks of active participation. In addition, there will be a 4-week, post-Taper completion follow-up for maximum total of 18-week trial duration
Description: All reports of a Serious Adverse Event (SAE) or an Unexpected Adverse Event (UAE) will be investigated by the monitoring team and reported to Washington University HRPO according to the reporting requirements.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/26
Other Adverse Events (participants affected / at risk) | 10/18 | 11/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=18) | Placebo (N=26)
fatigue (Investigations) | 10 (18) | 11 (26)
dizziness (Investigations) | 6 (18) | 0 (0)
weight gain (Investigations) | 5 (18) | 0 (0)
brain fog (Investigations) | 6 (18) | 2 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT05184192/Prot_SAP_000.pdf